CLINICAL TRIAL: NCT01782729
Title: The Efficacy and Safety of Tacrolimus Ointment in Pediatric Patients With Moderate to Severe Atopic Dermatitis
Brief Title: An Efficacy and Safety Study of Tacrolimus Ointment in Pediatric Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017827; R098924ADM4007
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, Atopic; Tacrolimus
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus ointment (pediatric) (Experimental): Tacrolimus ointment, 0.03 percent twice a day for pediatric population for 4 weeks or until 1 week after the affected areas defined for treatment at baseline are completely cleared, whichever is first.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus ointment, 0.03 percent twice a day for pediatric population for 4 weeks or until 1 week after the affected areas defined for treatment at baseline are completely cleared, whichever is first.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of tacrolimus ointment in treating the signs and symptoms of moderate (medium level of seriousness) to severe (very serious, life threatening) atopic dermatitis (an intensely pruritic [itching], chronic [lasting a long time], inflammatory [pain and swelling], immunologically based skin disease with a genetic predisposition [latent susceptibility to disease at the genetic level]) in pediatric participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) study in pediatric (2-12 years) participants with moderate to severe atopic dermatitis. Participants will be treated with 0.03 percent concentration of tacrolimus ointment which will be applied twice daily for 4 weeks or until 1 week after the affected areas defined for treatment at baseline are completely cleared, whichever is first. The study visits will consist of 6 visits: pre-study (optional), Baseline, Weeks 1, 2, 3 and 4. The ointment should be applied at least 2 hours before or at least 30 minutes after bathing, showering, shaving, use of sauna, or heavy exercise (i.e. causes sweating). On study visit days, the ointment should be applied at least 2 hours before the visit. Efficacy evaluation will be done at all subsequent study visits in participants receiving study drug for at least 3 consecutive days (minimum of 5 applications) while the participants who will receive at least 1 application of the study drug, will be evaluated for safety. Primary efficacy evaluation will be based on the Physician's Global Evaluation of Clinical Response (PhGECR). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion criteria :- Participants with a diagnosis of atopic dermatitis using Hanifin and Rajka Criteria (major criteria: pruritus, lichenification [crusting over], chronic relapsing [the return of a medical problem] course, family history of atopy and minor criteria: xerosis [dry skin], ichthyosis [skin disorders characterized by dryness, roughness, and scaliness], immediate Type I reactions [reactions which occur within minutes of exposure to challenging antigen: substances that are recognized by the immune system and induce an immune reaction] to skin test antigens) involving at least 10 percent of the body surface area

* Participants not having other skin disorders and severe heart, liver, kidney and lung diseases
* Participant or parent/guardian of pediatric participants has given informed consent
* Participants meets the following washout requirements (washout period ranging from 1 to 42 days) before the study: 1 day (for non-medicated topical [applied to skin; surface] agents); 7 days (for terfenadine, other non-sedating systemic antihistamines [drug used to treat allergic reaction], topical corticosteroids, H1 and H2 antihistamines, antimicrobial [drug that kills bacteria and other germs], other medicated topical agents); 14 days (for intranasal [delivery of medications through the nasal mucosa] and/or inhaled corticosteroids); 28 days (for light treatments [ultra violet rays A, ultra violet rays B], non-steroidal immunosuppressants [drug which suppresses the body's immune response, used in transplantation and diseases caused by disordered immunity], other investigational drugs and systemic corticosteroids); and 42 days (for astemizole)
* Participant and, if applicable, parent/guardian, agrees to comply with study requirements and is able to be at the clinic for all required study visits Exclusion Criteria: - Participants with a skin disorder other than atopic dermatitis in the treatment area
* Participant has pigmentation or extensive scarring or pigmented lesions (abnormal area of tissue, such as a wound, sore, rash, or boil) in the areas to be treated which would interfere with rating of efficacy parameters
* Participant has clinically infected atopic dermatitis at baseline
* Participants with a known hypersensitivity (altered reactivity to an antigen) to macrolides (drugs exhibiting antibiotic properties) or any excipient of the ointment
* Participant has a systemic disease, including cancer (abnormal tissue that grows and spreads in the body until it kills) or a history of cancer or Human Immunodeficiency Virus (HIV: a life-threatening infection which you can get from an infected person's blood or from having sex with an infected person), which would contraindicate (medical reasons that prevent a person from using a certain drug or treatment) the use of immunosuppressants

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Physician's Global Evaluation of Clinical Response (PhGECR) at Week 4 | Week 4
  The PhGECR scale evaluates the change in the lesions of atopic dermatitis, which is defined as the lesions identified by Investigator for treatment at Baseline only, using scores ranging from, less than 0 to 100: wherein, less than 0=worse, 0-29=no appreciable improvement, 30-49=slight improvement, 50-74=moderate improvement, 75-89=marked improvement, 90-99=excellent improvement and 100=cleared.

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Week 1, 2, 3 and 4
  A composite index of area involved and severity of the signs of atopic dermatitis in the 4 regions (head and neck, upper limbs, trunk, lower limbs) will be calculated using the physician's assessment of individual signs using a scale ranging from 0 to 3: 0=absent, 1=mild, 2=moderate, 3=severe; and the affected area assessment (the percentage of body surface area affected by atopic dermatitis) of the lesions defined in the baseline treatment area will be estimated by the physician on the basis of area score ranging from 0 to 6: 0=0 percent and 6=90 to 100 percent.
Participant's Assessment of Treatment Effects | Week 1, 2,3 and 4
  Participants will make two assessments at each study visit (before and after treatment) based on all affected areas (ratio of 100 percent). The assessment rates include: much better, better, slightly better, same, slightly worse, worse. Much better and better is considered good.
Participant's Assessment of Itch | Week 1,2, 3 and 4
  Participant's itch will be assessed using a Visual Analog Scale ranging from 0 to 100: 0-19=no or slight itch; 20-39=mild itch; 40-59=moderate itch; 60-79=severe itch; 80-100=worst itch.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (1):
- Hanoi, Vietnam

REFERENCES:
- See also: The efficacy and safety of tacrolimus ointment in pediatric patients with moderate to severe atopic dermatitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2485&filename=CR017827_CSR.pdf